CLINICAL TRIAL: NCT05146596
Title: The Effectiveness of Using Low-level Light Therapy to Treat Sleep and Psychological Symptoms Among Shift-work Nurses：A Randomized-controlled Trial
Brief Title: The Effectiveness of Using Low-level Light Therapy to Treat Sleep and Psychological Symptoms Among Shift-work Nurses
Acronym: t-PBM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-06-010C
Record Dates: First submitted 2021-07-29; First posted 2021-12-07 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Shift Work Type Circadian Rhythm Sleep Disorder
Keywords: Anxiety; Depression; nurses; LLLT
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: 1.Registered nurses who consciously have insomnia and ISI>=9. 2. People who have clear consciousness, can understand and agree to participate in this research. 3. Registered nurses who have been on shifts in the past six months. 4. Have the same type of shift within the four weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLLT group (Experimental): use low level light therapy,The Dr.Tai's energy cap
  Interventions: Device: use low level light therapy,The Dr.Tai's energy cap
- control group (No Intervention): routine care.

INTERVENTIONS:
Device: use low level light therapy,The Dr.Tai's energy cap — 30 minutes each time, three times a week, a total of 12 times.
  Arms: LLLT group

SUMMARY:
The purpose of this study is to explore the treatment of Low Level Light Therapy(LLLT) mitigate possible insomnia and psychological symptoms, when nurses have taken shifts.The investigators hope that the goal of this interventional research is to improve sleep quality and psychological symptoms of shift nurses in order to promote health.

DETAILED DESCRIPTION:
Low-Level Light Therapy; LLLT is also called PhotoBioModulation; PBM, which is a new type of interventional therapy.LLLT applies low-level lasers or light-emitting diodes(LEDs) to the human body for treatment. The wavelength of irradiated light is between red light(630-700 nm) and near-infrared light(700nm-1,100nm), and leads to a positive biological effect. It is a safe, painless, non-invasive treatment method. When LLLT is applied to the brain, it can pass through the scalp, head bone and reach the brain, and then stimulating the photochemical reaction in the cells, This is called transcranial Low-Level Laser Therapy (t-LLLT) or transcranial Photobiomodulation(t-PBM). tLLLT has existed since 1967, and more than thousands of scientific studies have shown that photons can stimulate biological responses and promote the normal work of cells. t-LLLT can treat a variety of diseases, such as emotional symptoms, lower back pain, weight loss, skin anti-aging, wound healing, etc. There are no reports of side effects. The main mechanism is similar to the photosynthesis of plants. It absorbs light and produces chemical reactions, supports mitochondrial function, and significantly increases the production of ATP(the main carrier of energy in cells.)in the brain, so as to function work better and achieve self-repair. This research uses Dr. Tai's energy cap, the manufacturer is Topunion Globaltek Inc., which passed the certification of the Ministry of Health and Welfare(MOHW) for medical device in 2019. It has been modified to the second generation and is now on the market. It basically provides two kinds of red light (wavelength of 660nm) and near-infrared light(wavelength of 850nm), which is mainly used at home. The research intervention will be conducted for four weeks, pre-tests and post-tests will be conducted as indicators to evaluating sleep and psychological symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Registered nurses who consciously have insomnia and ISI>=9.
2. People who have clear consciousness, can understand and agree to participate in this research.
3. Registered nurses who have been on shifts in the past six months.
4. Have the same type of shift within the four weeks.

Exclusion Criteria:

1. Those who have undergone head surgery.
2. Those who are pregnant.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
psychological symptoms | 1 month,up to 4 weeks.measure every 1 week.Change from baseline DASS-21 at 1,2,3,4 weeks, a total of five times.
  use scale:Depression Anxiety Stress Scale-21(DASS-21)measure psychological symptoms.There are a total of 21 questions on the scale, each with a score of 3 and a score of 0 to 63. The higher score mean a worse outcome,mean psychological symptoms are severe.The higher the score the more severe the symptoms, the lower the score the more minor.

SECONDARY OUTCOMES:
sleep symptoms | 1 month,up to 4 weeks.Change from baseline ISI at 2,4 weeks.
  use scale:Insomnia Severity Index(ISI) measure sleep symptoms.There are a total of 7 questions on the scale, each with a score of 4 and a score of 0 to 28. The higher score mean a worse outcome,mean sleep symptoms are severe.The study measure use ISI scale every 2 weeks
instrument:Heart rate variability(HRV) | Measure three days a week, two time points (T0, T1) for each measurement, T0=baseline, and T1=after 30mins,24 times in both groups.
  heart rhythm variability and autonomic nerves, so this study used this instrument as an objective data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Liao General Y Hsuan, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Liao General Yung Hsuan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The research is in progress and will not be published until it is completed.

REFERENCES:
- [Result] Hamblin MR. Photobiomodulation or low-level laser therapy. J Biophotonics. 2016 Dec;9(11-12):1122-1124. doi: 10.1002/jbio.201670113. No abstract available. PMID 27973730
- [Derived] Liao YH, Tai CJ, Ming JL, Lin LH, Chien LY. The Effectiveness of Low-Level LED Light Therapy for Sleep Problems, Psychological Symptoms, and Heart Rate Variability in Shift-Work Nurses: A Randomized Controlled Trial. J Nurs Manag. 2025 Jun 17;2025:6478834. doi: 10.1155/jonm/6478834. eCollection 2025. PMID 40557249
- See also: Photobiomodulation or low-level laser therapy — http://onlinelibrary.wiley.com/doi/10.1002/jbio.201670113